CLINICAL TRIAL: NCT06541405
Title: An Open, Single Center Exploratory Study to Evaluate Safety and Efficacy of NK520 for Pediatric Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Safety and Efficacy of NK520 to Treat Pediatric Relapsed/Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Base Therapeutics (Shanghai) Co., Ltd. (Industry)
Collaborators: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NK520-01
Record Dates: First submitted 2024-06-07; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-05

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A(low-dose group) (Experimental): NK520: 5x10^7 NK/kg
  Interventions: Drug: NK520
- Group B(medium-dose group) (Experimental): NK520: 1.5×10^8NK/kg
  Interventions: Drug: NK520
- Group C(high-dose group) (Experimental): NK520: 3×10^8NK/kg
  Interventions: Drug: NK520

INTERVENTIONS:
Drug: NK520 — The number of NK520 cell infused for each dosing should be calculated base on the body weight of subject. NK520 will be administered through intravenous infusion.
  Other Names: genetic modified NK cell

SUMMARY:
This study will evaluate the safety and efficacy of NK520 in the treatment of pediatric relapsed/refractory acute myeloid leukemia. NK520 will be administered by intravenous injection. The safety and efficacy of this treatment will be evaluated.

DETAILED DESCRIPTION:
This open label, single-arm study aims to evaluate the efficacy and safety of allogenic NK cells in pediatric relapsed/refractory acute myeloid leukemia. Allogenic NK cells will be infused once a week. After infusion, the investigators will observe the characteristics of dose limited toxicity (DLT), and determine the maximum tolerable dose(MTD). To provide basis for the dosage and treatment plan of cell products in follow-up clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be between 6 and 18 years;
2. Diagnostic Criteria: Meet the 2022 World Health Organization (WHO) diagnostic criteria for AML, unsuitable for current treatments or patients with relapsed/refractory AML after ≥2 lines of therapy. The definition of relapsed/refractory acute myeloid leukemia is based on the 2017 Chinese Guidelines for Diagnosis and Treatment: a. Relapsed AML: Diagnosis is confirmed when leukemia cells reappear in the peripheral blood or bone marrow blast cells exceed 5% after complete remission (CR) (excluding reasons such as bone marrow regeneration post-consolidation chemotherapy) or there is extramedullary infiltration by leukemia cells; b. Refractory AML: Initial cases unresponsive after two cycles of standard regimen treatment; recurrence within 12 months after CR and consolidation therapy; recurrence beyond 12 months with ineffectiveness of conventional chemotherapy; those who have relapsed twice or more; or persistent extramedullary leukemia;
3. For participants under 16 years old, Lansky performance status must be ≥50%; for participants aged 16 or older, Karnofsky performance status must be ≥50%;
4. Expected survival of at least 12 weeks;
5. Normal Organ Function.

Exclusion Criteria:

1. Acute promyelocytic leukemia, chronic myeloid leukemia, acute mixed lineage leukemia, or known central nervous system leukemia;
2. AML associated with congenital syndromes, such as Down syndrome, Fanconi anemia, Bloom syndrome, Kostmann syndrome, or congenital aplastic anemia;
3. Severe bleeding tendency or coagulation disorders, or currently receiving thrombolytic therapy;
4. HIV-infected individuals, or individuals with known active syphilis infection;
5. Receipt of live attenuated vaccines within 2 weeks before the first dose or planned during the study period;
6. Participation in another clinical trial and receipt of investigational drug within 4 weeks prior to the first dose;
7. Receipt of immune-modulatory drugs (including thymosin, interferons, except for local use to manage conditions like pleural or ascites fluid) within 2 weeks before the first dose;
8. At screening, positive hepatitis B or C viral markers as follows:

   * HBsAg positive with serum HBV-DNA level ≥1×10^3 copies/mL or above normal range;
   * Positive for HCV antibodies;
9. Any other condition or situation in which the investigator deems the patient unsuitable for participation in this study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity | From the first infusion of NK520 to 4 weeks after last infusion of NK520
  To evaluate the DLT during N520 treatment
Complete Response Rate (CRR) | from the date of first infusion of NK510 up to 104 weeks
  Effectiveness Metrics

SECONDARY OUTCOMES:
Overall response rate (ORR) | from the date of first infusion of NK510 up to 104 weeks
  Effectiveness Metrics
Duration of Response (DOR) | From the date of enrollment up to 104 weeks
  Effectiveness Metrics
Event-Free Survival (EFS) | From date of enrollment up to 104 weeks, or progression, or date of death, whichever came first.
  Effectiveness Metrics
Overall Survival (OS) | From date of enrollment up to 104 weeks, or date of death, whichever came first.
  Effectiveness Metrics

CONTACTS AND LOCATIONS:
Overall Officials: wenting Hu, Principal Investigator — Shanghai children's medical center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No